CLINICAL TRIAL: NCT01716520
Title: A Randomized, Double-Blind, 3-Way, Cross-Over Study to Evaluate Lung Function Response After Treatment With Umeclidinium 62.5mcg, Vilanterol 25mcg, and Umeclidinium/Vilanterol 62.5/25mcg Once-Daily in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Cross-Over Study in Subjects With COPD, Evaluating Lung Function Response After Treatment With Once Daily Umeclidinium 62.5mcg, Vilanterol 25mcg, and Umeclidinium/Vilanterol 62.5/25mcg
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 116133
Record Dates: First submitted 2012-10-11; First posted 2012-10-30 (Estimated); Results first posted 2014-02-11 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: long-acting muscarinic antagonist; long-acting beta-agonist; Chronic Obstructive Pulmonary Disease; vilanterol; umeclidinium
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Umeclidinium/Vilanterol 62.5/25 mcg (Experimental): Umeclidinium/Vilanterol 62.5/25 mcg once daily in the morning via novel dry powder inhaler (NDPI)
  Interventions: Device: Umeclidinium/Vilanterol 62.5/25 mcg
- Umeclidinium 62.5 mcg (Experimental): Umeclidinium 62.5 mcg once daily in the morning via novel dry powder inhaler (NDPI)
  Interventions: Device: Umeclidinium 62.5 mcg
- Vilanterol 25 mcg (Experimental): Vilanterol 25 mcg once daily in the morning via novel dry powder inhaler (NDPI)
  Interventions: Device: Vilanterol 25 mcg

INTERVENTIONS:
Device: Umeclidinium/Vilanterol 62.5/25 mcg — Umeclidinium/Vilanterol 62.5/25 mcg once daily in the morning via novel dry powder inhaler (NDPI)
  Arms: Umeclidinium/Vilanterol 62.5/25 mcg
Device: Umeclidinium 62.5 mcg — Umeclidinium 62.5 mcg once daily in the morning via novel dry powder inhaler (NDPI)
  Arms: Umeclidinium 62.5 mcg
Device: Vilanterol 25 mcg — Vilanterol 25 mcg once daily in the morning via novel dry powder inhaler (NDPI)
  Arms: Vilanterol 25 mcg

SUMMARY:
The purpose of this study is to evaluate the lung function response to UMEC/VI, UMEC, and VI in individual patients using a cross-over design. This is a multicenter, randomized, double-blind, 3-way crossover study. Eligible subjects will be randomized to a sequence of UMEC 62.5mcg, VI 25mcg, and UMEC/VI 62.5/25mcg. All subjects will receive each treatment once-daily for 14 days, and each treatment will be separated by a 10-14 day washout period. There will be a 5-7 day run-in period prior to randomization.

ELIGIBILITY:
Inclusion Criteria:

* Type of Patient: Outpatient
* Informed Consent: A signed and dated written informed consent prior to study participation
* Age: Subjects 40 years of age or older at Visit 1
* Gender: Male or female subjects.
* COPD diagnosis: As defined by the American Thoracic Society/European Respiratory Society (ATS/ERS)
* Severity of disease: A pre- and post-salbutamol FEV1/FVC ratio of <0.70 and a pre- and post-salbutamol FEV1 of ≤ 70% of predicted normal values at Visit 1
* Smoking History: Current or former cigarette smokers with a history of cigarette smoking of ≥ 10 pack-years at Visit 1
* Female subject of non child-bearing potential OR a female subject of child bearing potential, with a negative pregnancy test at screening, and agreeing to consistently and correctly use one of the acceptable contraceptive methods

Exclusion Criteria:

* Pregnancy: Women who are pregnant or lactating or are planning on becoming pregnant during the study
* Asthma: A current diagnosis of asthma
* Other Respiratory Disorders: Known alpha-1 antitrypsin deficiency, active lung infections (such as tuberculosis), and lung cancer are absolute exclusionary conditions.
* Other Diseases/Abnormalities: Subjects with historical or current evidence of clinically significant cardiovascular, neurological, psychiatric, renal, hepatic, immunological, endocrine (including uncontrolled diabetes or thyroid disease) or hematological abnormalities that are uncontrolled and/or a previous history of cancer in remission for < 5 years prior to Visit 1
* Contraindications: A history of allergy or hypersensitivity to any anticholinergic/muscarinic receptor antagonist, beta2-agonist, lactose/milk protein or magnesium stearate or a medical condition such as of narrow-angle glaucoma, prostatic hypertrophy or bladder neck obstruction that, in the opinion of the study physician contraindicates study participation or use of an inhaled anticholinergic.
* Hospitalization: Hospitalization for COPD or pneumonia within 12 weeks prior to Visit 1.
* Lung Resection: Subjects with lung volume reduction surgery within the 12 months prior to Visit 1.
* 12-Lead ECG: An abnormal and significant ECG finding from the 12-lead ECG conducted at Visit 1
* Screening Labs: Significantly abnormal finding from clinical chemistry or hematology tests at Visit 1 as determined by the study investigator.
* Medication Prior to Spirometry: Unable to withhold salbutamol for the 4 hour period required prior to spirometry testing at each study visit and at each spirometry test performed at home.
* Medications Prior to Screening: Use of the prohibited medications according to defined time intervals prior to Visit 1
* Oxygen: Use of long-term oxygen therapy (LTOT) described as oxygen therapy prescribed for greater than 12 hours a day. As-needed oxygen use (i.e., ≤ 12 hours per day) is not exclusionary.
* Nebulized Therapy: Regular use (prescribed for use every day, not for as-needed use) of short-acting bronchodilators (e.g., salbutamol, ipratropium bromide) via nebulized therapy
* Pulmonary Rehabilitation Program: Participation in the acute phase of a pulmonary rehabilitation program within 4 weeks prior to Visit 1. Subjects who are in the maintenance phase of a pulmonary rehabilitation program are not excluded.
* Drug or Alcohol Abuse: A known or suspected history of alcohol or drug abuse within 2 years prior to Visit 1.
* Affiliation with Investigator Site: Is an investigator, sub-investigator, study coordinator, employee of a participating investigator or study site, or immediate family member of the aforementioned that is involved in this study.
* Inability to read: In the opinion of the Investigator, any subject who is unable to read and/or would not be able to complete a questionnaire

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2012-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (16):
- Estonia (3):
  - GSK Investigational Site, Haapsalu
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Germany (13):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Nuremberg, Bavaria
  - GSK Investigational Site, Potsdam, Brandenburg
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Rodgau, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzg, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Großhansdorf, Schleswig-Holstein
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 116133 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116133 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116133 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116133 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116133 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116133 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116133 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who met the eligibility criteria at screening (Visit 1) completed a 5- to 7-day run-in period prior to being randomized to 1 of 6 treatment sequences. The treatment phase was comprised of three 14-day treatment periods, each separated by a 10- to 14-day washout period, starting on Day 15.
Groups:
- Sequence 1: UMEC 62.5 µg, VI 25 µg, UMEC/VI 62.5/25 µg: Participants received umeclidinium (UMEC) 62.5 micrograms (µg), vilanterol (VI) 25 µg, and UMEC/VI 62.5/25 µg in Treatment Periods 1, 2, and 3, respectively. Participants received all treatments once a day (QD) for 14 days from a Dry Powder Inhaler (DPI). The three treatment periods were separated by a washout period of 10 to 14 days.
- Sequence 2: VI 25 µg, UMEC/VI 62.5/25 µg, UMEC 62.5 µg: Participants received VI 25 µg, UMEC/VI 62.5/25 µg, and UMEC 62.5 µg in Treatment Periods 1, 2, and 3, respectively. Participants received all treatments QD for 14 days from a DPI. The three treatment periods were separated by a washout period of 10 to 14 days.
- Sequence 3: UMEC/VI 62.5/25 µg, UMEC 62.5 µg, VI 25 µg: Participants received UMEC/VI 62.5/25 µg, UMEC 62.5 µg, and VI 25 µg in Treatment Periods 1, 2, and 3, respectively. Participants received all treatments QD for 14 days from a DPI. The three treatment periods were separated by a washout period of 10 to 14 days.
- Sequence 4: UMEC 62.5 µg, UMEC/VI 62.5/25 µg, VI 25 µg: Participants received UMEC 62.5 µg, UMEC/VI 62.5/25 µg, and VI 25 µg in Treatment Periods 1, 2, and 3, respectively. Participants received all treatments QD for 14 days from a DPI. The three treatment periods were separated by a washout period of 10 to 14 days.
- Sequence 5: VI 25 µg, UMEC 62.5 µg, UMEC/VI 62.5/25 µg: Participants received VI 25 µg, UMEC 62.5 µg, and UMEC/VI 62.5/25 µg in Treatment Periods 1, 2, and 3, respectively. Participants received all treatments QD for 14 days from a DPI. The three treatment periods were separated by a washout period of 10 to 14 days.
- Sequence 6: UMEC/VI 62.5/25 µg, VI 25 µg, UMEC 62.5 µg: Participants received UMEC/VI 62.5/25 µg, VI 25 µg, and UMEC 62.5 µg in Treatment Periods 1, 2, and 3, respectively. Participants received all treatments QD for 14 days from a DPI. The three treatment periods were separated by a washout period of 10 to 14 days.
Period: Treatment Period 1 (14 Days)
Arm/Group | Sequence 1: UMEC 62.5 µg, VI 25 µg, UMEC/VI 62.5/25 µg | Sequence 2: VI 25 µg, UMEC/VI 62.5/25 µg, UMEC 62.5 µg | Sequence 3: UMEC/VI 62.5/25 µg, UMEC 62.5 µg, VI 25 µg | Sequence 4: UMEC 62.5 µg, UMEC/VI 62.5/25 µg, VI 25 µg | Sequence 5: VI 25 µg, UMEC 62.5 µg, UMEC/VI 62.5/25 µg | Sequence 6: UMEC/VI 62.5/25 µg, VI 25 µg, UMEC 62.5 µg
Started | 31 | 30 | 30 | 30 | 31 | 30
Completed | 29 | 29 | 28 | 29 | 31 | 29
Not Completed | 2 | 1 | 2 | 1 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol-defined Stopping Criteria | 1 | 0 | 2 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Period: Washout Period 1 (10 to 14 Days)
Arm/Group | Sequence 1: UMEC 62.5 µg, VI 25 µg, UMEC/VI 62.5/25 µg | Sequence 2: VI 25 µg, UMEC/VI 62.5/25 µg, UMEC 62.5 µg | Sequence 3: UMEC/VI 62.5/25 µg, UMEC 62.5 µg, VI 25 µg | Sequence 4: UMEC 62.5 µg, UMEC/VI 62.5/25 µg, VI 25 µg | Sequence 5: VI 25 µg, UMEC 62.5 µg, UMEC/VI 62.5/25 µg | Sequence 6: UMEC/VI 62.5/25 µg, VI 25 µg, UMEC 62.5 µg
Started | 29 | 29 | 28 | 29 | 31 | 29
Completed | 29 | 28 | 27 | 29 | 31 | 27
Not Completed | 0 | 1 | 1 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 1
Period: Treatment Period 2 (14 Days)
Arm/Group | Sequence 1: UMEC 62.5 µg, VI 25 µg, UMEC/VI 62.5/25 µg | Sequence 2: VI 25 µg, UMEC/VI 62.5/25 µg, UMEC 62.5 µg | Sequence 3: UMEC/VI 62.5/25 µg, UMEC 62.5 µg, VI 25 µg | Sequence 4: UMEC 62.5 µg, UMEC/VI 62.5/25 µg, VI 25 µg | Sequence 5: VI 25 µg, UMEC 62.5 µg, UMEC/VI 62.5/25 µg | Sequence 6: UMEC/VI 62.5/25 µg, VI 25 µg, UMEC 62.5 µg
Started | 29 | 28 | 27 | 29 | 31 | 27
Completed | 29 | 28 | 27 | 28 | 29 | 27
Not Completed | 0 | 0 | 0 | 1 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol-defined Stopping Criteria | 0 | 0 | 0 | 1 | 0 | 0
Period: Washout Period 2 (10 to 14 Days)
Arm/Group | Sequence 1: UMEC 62.5 µg, VI 25 µg, UMEC/VI 62.5/25 µg | Sequence 2: VI 25 µg, UMEC/VI 62.5/25 µg, UMEC 62.5 µg | Sequence 3: UMEC/VI 62.5/25 µg, UMEC 62.5 µg, VI 25 µg | Sequence 4: UMEC 62.5 µg, UMEC/VI 62.5/25 µg, VI 25 µg | Sequence 5: VI 25 µg, UMEC 62.5 µg, UMEC/VI 62.5/25 µg | Sequence 6: UMEC/VI 62.5/25 µg, VI 25 µg, UMEC 62.5 µg
Started | 29 | 28 | 27 | 28 | 29 | 27
Completed | 27 | 27 | 26 | 28 | 29 | 25
Not Completed | 2 | 1 | 1 | 0 | 0 | 2
Not completed — Adverse Event | 1 | 0 | 1 | 0 | 0 | 1
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol-defined Stopping Criteria | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Period: Treatment Period 3 (14 Days)
Arm/Group | Sequence 1: UMEC 62.5 µg, VI 25 µg, UMEC/VI 62.5/25 µg | Sequence 2: VI 25 µg, UMEC/VI 62.5/25 µg, UMEC 62.5 µg | Sequence 3: UMEC/VI 62.5/25 µg, UMEC 62.5 µg, VI 25 µg | Sequence 4: UMEC 62.5 µg, UMEC/VI 62.5/25 µg, VI 25 µg | Sequence 5: VI 25 µg, UMEC 62.5 µg, UMEC/VI 62.5/25 µg | Sequence 6: UMEC/VI 62.5/25 µg, VI 25 µg, UMEC 62.5 µg
Started | 27 | 27 | 26 | 28 | 29 | 25
Completed | 27 | 27 | 25 | 28 | 29 | 23
Not Completed | 0 | 0 | 1 | 0 | 0 | 2
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- UMEC 62.5 µg, VI 25 µg, UMEC/VI 62.5/25 µg: All participants received one of the following three treatments in one of three treatment periods QD from the DPI for 14 days: UMEC 62.5 µg inhalation powder; VI 25 µg inhalation powder; and UMEC/VI 62.5/25 µg inhalation powder. Participants were randomized to receive treatment in one of the six following sequences: (1) UMEC 62.5 µg, VI 25 µg, UMEC/VI 62.5/25 µg; (2) VI 25 µg, UMEC/VI 62.5/25 µg, UMEC 62.5 µg; (3) UMEC/VI 62.5/25 µg, UMEC 62.5 µg, VI 25 µg; (4) UMEC 62.5 µg, UMEC/VI 62.5/25 µg, VI 25 µg; (5) VI 25 µg, UMEC 62.5 µg, UMEC/VI 62.5/25 µg; (6) UMEC/VI 62.5/25 µg, VI 25 µg, UMEC 62.5 µg. The three treatment periods were separated by a washout period of 10 to 14 days.
Arm/Group | UMEC 62.5 µg, VI 25 µg, UMEC/VI 62.5/25 µg
Number analyzed (Participants) | 182
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.2 (8.19)
Gender [Count of Participants; unit: Participants]
  Female | 55
  Male | 127
Race/Ethnicity, Customized [Number; unit: participants]
  White - White/Caucasian/European Heritage | 182

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (BL) in Weighted Mean (WM) 0-6 Hour Forced Expiratory Volume in One Second (FEV1) Obtained Post-dose at Day 14 of Each Treatment Period (TP) by Response Type
Description: FEV1 is a measure of lung function and the maximal amount of air that can be forcefully exhaled in one second. The WM FEV1 was derived by calculating the area under the FEV1/time curve (AUC) using the trapezoidal rule, and then dividing the value by the time interval over which the AUC was calculated. The WM FEV1 was calculated using 0-6 hour post-dose measurements at Day 14 of each TP, which included pre-dose (trough value for Day 14 [mean of the 23 and 24 hour assessments post Day 13 dosing]) and post-dose 15 minutes (min), 30 min, and 1, 3, and 6 hours. BL is the mean FEV1 values recorded 30 min and 5 min pre-dose on Day 1 of each TP, mean BL is the mean of the BLs for each participant, and period BL is the difference between the BL and the mean BL in each TP for each participant. Change from BL for each TP is the Day 14 value minus the BL value for that TP. Participants could have been classified as responders to both UMEC and VI.
Time Frame: Baseline and Day 14 of each treatment period (up to study day 83)
Population: Intent-to-Treat (ITT) Population: all participants (par.) randomized to treatment who received >=1 dose of randomized study medication in a TP. Only par. available at the specified time points were analyzed. Different par. may have been analyzed for different parameters; the overall number of par, analyzed reflects everyone in the ITT Population.
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- UMEC 62.5 µg: Participants received UMEC 62.5 µg inhalation powder QD from the DPI for 14 days during one of the three treatment periods. Each treatment period was followed by a washout period of 10-14 days.
- VI 25 µg: Participants received VI 25 µg inhalation powder QD from the DPI for 14 days during one of the three treatment periods. Each treatment period was followed by a washout period of 10-14 days.
- UMEC/VI 62.5/25 µg: Participants received UMEC/VI 62.5/25 µg inhalation powder QD from the DPI for 14 days during one of the three treatment periods. Each treatment period was followed by a washout period of 10-14 days.
Arm/Group | UMEC 62.5 µg | VI 25 µg | UMEC/VI 62.5/25 µg
Number analyzed (Participants) | 171 | 171 | 173
Liters
  Responder to UMEC, n=90, 90, 88 | 0.216 (0.0166) | 0.201 (0.0167) | 0.337 (0.0166)
  Responder to VI, n=99, 102, 100 | 0.189 (0.0150) | 0.233 (0.0147) | 0.331 (0.0148)
  Responder to Neither, n=36, 37, 36 | 0.077 (0.0243) | 0.057 (0.0240) | 0.130 (0.0243)
Statistical Analysis 1: Comparison: UMEC 62.5 µg vs UMEC/VI 62.5/25 µg; Test type: Superiority or Other; p < 0.001, ANCOVA — Analysis was performed using an Analysis of Covariance (ANCOVA) model with covariates of treatment, period, mean Baseline, period Baseline, response type and treatment by response type interaction; Mean Difference (Final Values) = 0.121, 95% CI 2-sided [0.085 to 0.157] — Responders to UMEC=responders to UMEC or to both monotherapies, as defined by a participant with an increase from Baseline of >=12% and 200 milliliters (mL) at >=1 time point over 0-6 hours post-dose in FEV1 on Day 1
Statistical Analysis 2: Comparison: VI 25 µg vs UMEC/VI 62.5/25 µg; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.135, 95% CI 2-sided [0.100 to 0.171] — Responders to UMEC=responders to UMEC or to both monotherapies, as defined by a participant with an increase from Baseline of >=12% and 200 mL at >=1 time point over 0-6 hours post-dose in FEV1 on Day 1
Statistical Analysis 3: Comparison: UMEC 62.5 µg vs UMEC/VI 62.5/25 µg; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.142, 95% CI 2-sided [0.110 to 0.174] — Responders to VI=responders to VI or to both monotherapies, as defined by a participant with an increase from Baseline of >=12% and 200 mL at >=1 time point over 0-6 hours post-dose in FEV1 on Day 1
Statistical Analysis 4: Comparison: VI 25 µg vs UMEC/VI 62.5/25 µg; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.098, 95% CI 2-sided [0.067 to 0.130] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 5: Comparison: UMEC 62.5 µg vs UMEC/VI 62.5/25 µg; Test type: Superiority or Other; p = 0.047, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.052, 95% CI 2-sided [0.001 to 0.104] — Responders to Neither=responders to neither UMEC nor VI, as defined by a participant with at least one FEV1 assessment over 0-6 hours post-dose on Day 1 but no increase from Baseline of >=12% and 200 mL at any assessment(s)
Statistical Analysis 6: Comparison: VI 25 µg vs UMEC/VI 62.5/25 µg; Test type: Superiority or Other; p = 0.006, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.073, 95% CI 2-sided [0.021 to 0.124] — [estimate comment as in outcome 1, analysis 5]

2. Secondary Outcome: Number of Participants (Par.) Who Were Responsive to UMEC/VI, UMEC, or VI According to FEV1 at Day 1 of Each Treatment Period (TP)
Description: A responder is a par. with an increase from BL of >=12% and 200 milliliters (mL) at >=1 time point over 0-6 hours post-dose (PD) in FEV1 on Day 1. A non-responder (NR) is a par. with >=1 FEV1 assessment over 0-6 hours PD on Day 1 but no increase from BL of >=12% and 200 mL at any assessment(s). Missing: no FEV1 data recorded over 0-6 hours PD on Day 1. Response type is defined based on a par.'s response to each individual monotherapy treatment. A responder to UMEC is a par. who is a responder in the UMEC treatment period (TP) and either a NR or has missing data in the VI TP. A responder to VI is a par. who is a responder in the VI TP and either a NR or has missing data in the UMEC TP. A responder to UMEC and VI is a par. who is a responder in both the UMEC and VI TPs. A responder to neither is a par. who is a NR in both the UMEC and VI TPs. Missing: a par. who has missing data in both the UMEC and VI TPs, or who has missing data in one monotherapy period and is a NR in the other.
Time Frame: Baseline (BL) and 0-6 hours post-dose (15 minutes, 30 minutes, and 1, 3, and 6 hours post-dose) on Day 1 of each treatment period (up to study day 71)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | UMEC 62.5 µg | VI 25 µg | UMEC/VI 62.5/25 µg
Number analyzed (Participants) | 171 | 171 | 173
participants
  Responders | 92 | 104 | 124
  Non-responders | 79 | 67 | 49

3. Secondary Outcome: Number of Participants With a Larger Change From Baseline in 0-6 Hour Weighted Mean FEV1 at Day 14 of Each Treatment Period With UMEC/VI Compared With UMEC and VI Alone
Description: The number of participants with a larger change from Baseline in weighted mean FEV1 with UMEC/VI compared with UMEC and VI alone was recorded. Participants who improved on UMEC/VI had a larger change from Baseline difference in 0-6 hour weighted mean FEV1 on Day 14 on UMEC/VI compared to UMEC or VI alone. Baseline is the mean FEV1 values recorded 30 min and 5 min pre-dose on Day 1 of each treatment period, mean Baseline is the mean of the Baselines for each participant, and period Baseline is the difference between the Baseline and the mean Baseline in each treatment period for each participant. Change from Baseline for each treatment period is the Day 14 value minus the Baseline value for that treatment period.
Time Frame: Baseline and Day 14 of each treatment period (up to study day 83)
Population: ITT Population. Only those participants available at the specified time point were analyzed.
Measure: Number; unit: participants
Arm/Group | UMEC 62.5 µg | VI 25 µg
Number analyzed (Participants) | 162 | 163
participants
  Improved on UMEC/VI | 113 | 121
  Not Improved on UMEC/VI | 49 | 42

4. Secondary Outcome: Change From Baseline in Trough FEV1 on Day 15 of Each Treatment Period
Description: Trough FEV1 on Treatment Day 15 is defined as the mean of the FEV1 values obtained at 23 and 24 hours after dosing on Day 14. Analysis was performed using an ANCOVA model with covariates of treatment, period, mean Baseline (BL), period BL, response type, and treatment by response type interaction. A participant is a reponder to UMEC if they were a responder to UMEC monotherapy or a responder to both UMEC monotherapy and VI monotherapy. A participant is a responder to VI if they were a responder to VI monotherapy or a responder to both UMEC monotherapy or VI monotherapy. BL is the mean FEV1 recorded 30 min and 5 min pre-dose on Day 1 of each treatment period, mean BL is the mean of the BLs for each participant, and period BL is the difference between BL and the mean BL in each treatment period for each participant. Change from BL for each treatment period is the Day 15 value minus the BL value for that treatment period.
Time Frame: Baseline and Day 15 of each treatment period (up to study day 84)
Population: ITT Population. Only those participants available at the specified time points were analyzed. Different participants may have been analyzed for different parameters; the overall number of participants analyzed reflects everyone in the ITT Population.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | UMEC 62.5 µg | VI 25 µg | UMEC/VI 62.5/25 µg
Number analyzed (Participants) | 171 | 171 | 173
Liters
  Responder to UMEC, n=90, 89, 87 | 0.159 (0.0178) | 0.134 (0.0180) | 0.242 (0.0179)
  Responder to VI, n=99, 101, 99 | 0.135 (0.0160) | 0.161 (0.0158) | 0.268 (0.0159)
  Responder to Neither, n=35, 37, 36 | 0.060 (0.0263) | 0.035 (0.0257) | 0.092 (0.0260)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of study medication to the end of the treatment period (up to Study Week 12).
Description: SAEs and non-serious AEs were reported for members of the Intent-to-Treat (ITT) Population, comprised of all participants randomized to treatment who received at least one dose of trial medication during the treatment period.
Arm/Group | UMEC 62.5 µg | VI 25 µg | UMEC/VI 62.5/25 µg
Serious Adverse Events (participants affected / at risk) | 3/171 | 1/171 | 3/173
Other Adverse Events (participants affected / at risk) | 8/171 | 13/171 | 13/173
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UMEC 62.5 µg (N=171) | VI 25 µg (N=171) | UMEC/VI 62.5/25 µg (N=173)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Abscess limb (Infections and infestations) | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | UMEC 62.5 µg (N=171) | VI 25 µg (N=171) | UMEC/VI 62.5/25 µg (N=173)
Nasopharyngitis (Infections and infestations) | 5 | 11 | 7
Headache (Nervous system disorders) | 3 | 2 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.